CLINICAL TRIAL: NCT05370326
Title: Randomized Controlled Pilot Trial to Evaluate Feasibility and Preliminary Efficacy of an Opioid Stewardship Program in Hospitalized Patients With Chronic Pain
Brief Title: Feasibility and Preliminary Efficacy of an Opioid Stewardship Program in Hospitalized Patients With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2000032638; 1RM1DA055310-01 (NIH)
Record Dates: First submitted 2022-05-04; First posted 2022-05-11 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Opioid Dependence; Chronic Pain
MeSH Terms: conditions — Opioid-Related Disorders; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Opioid Stewardship Program (Experimental): Enhanced opioid stewardship program, tailored to the needs of hospitalized patients with chronic pain with opioid dependence, incorporating real-time guidance from an addiction medicine and pain-trained physician/pharmacist team
  Interventions: Other: Enhanced Opioid Stewardship Program
- Standard of care (No Intervention)

INTERVENTIONS:
Other: Enhanced Opioid Stewardship Program — The goal of the enhanced opioid stewardship intervention is to manage chronic pain while reducing risk of inappropriate/risky opioid use and preventing harms of opioid use.
  Arms: Enhanced Opioid Stewardship Program

SUMMARY:
This study aims to investigate the feasibility and preliminary efficacy of an enhanced opioid stewardship program, tailored to the needs of hospitalized patients with chronic pain with opioid dependence, incorporating real-time guidance from an addiction medicine and pain-trained physician/pharmacist team, using a pilot randomized clinical trial format. Findings from this research may improve pain management and decrease risk of opioid-related adverse events among patients with chronic pain.

DETAILED DESCRIPTION:
The primary objective of this study is to determine whether an enhanced opioid stewardship program, tailored to the needs of patients with chronic pain, is feasible to implement in a hospital setting.

One secondary objective is to determine whether an enhanced opioid stewardship program increases use of guideline-based opioid care. The other secondary objective of this study is to determine whether an enhanced opioid stewardship program reduces pain frequency, intensity, and interference and decreases the risk for opioid-related adverse events among adult patients with chronic pain hospitalized on medical units at Yale-New Haven Hospital, York Street and Saint Raphael campuses.

This is a pilot randomized controlled trial of 100 adult participants. It is prospective and focus primarily on feasibility. There will be up to 3 study visits with each participant, which will take place during hospitalization or in the first week after hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* admitted at Yale New Haven Hospital (YSC and SRC) on medical units
* identified as having chronic pain and prescribed opioids
* have opioid dependence (evidenced by ongoing opioid prescription, meeting Diagnostic and Statistical Manual of Mental Disorders-5 criteria for Opioid Use Disorder, or clinical history)

Exclusion Criteria:

* active cancer
* current pregnancy
* hospice care/comfort measures only
* admission to inpatient psychiatry
* completed or planned Addiction Medicine consult during hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Weimer, DO, MCR, FASAM, Principal Investigator — Yale University; Alexandra Hajduk, PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale New Haven Hospital, 20 York Street, New Haven, Connecticut
  - Yale New Haven Hospital, 1450 Chapel Street, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care: Participants received standard of care services without the enhanced opioid stewardship program.
Period: Overall Study
Arm/Group | Enhanced Opioid Stewardship Program | Standard of Care
Started | 36 | 16
Complete Clinical Data | 36 | 16
Complete Self Report Data | 31 | 14
Completed | 36 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants randomized in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Opioid Stewardship Program | Standard of Care | Total
Number analyzed (Participants) | 36 | 16 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (13.7) | 52.3 (15.0) | 53.7 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 10 | 28
  Male | 18 | 6 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 11
  Not Hispanic or Latino | 31 | 10 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 4 | 19
  White | 20 | 9 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 36 | 16 | 52

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Screened Compared to Number of Eligible Participants to Determine Feasibility of Recruitment
Description: Feasibility of recruitment will be determined by a count of the number of participants screened for the study compared to number of eligible participants.
Time Frame: approximately 3 months
Population: All participants that were screened for eligibility
Measure: Count of Participants; unit: Participants
Groups:
- Total Participants Screened: This is the total number of participants that were screened for eligibility.
Arm/Group | Total Participants Screened
Number analyzed (Participants) | 510
Participants
  Eligible participants approached | 97
  Ineligible participants due to Inclusion | 62
  Ineligible participants due to Exclusion | 351

2. Primary Outcome: Number of Eligible Participants Compared to Number of Enrolled Participants to Determine Feasibility of Recruitment
Description: Feasibility of recruitment will be determined by a count of the number of participants eligible for the study compared to number of enrolled participants.
Time Frame: approximately 3 months
Population: Total number of eligible participants.
Measure: Count of Participants; unit: Participants
Groups:
- Total Eligible Participants: The total number of participants found eligible for the study.
Arm/Group | Total Eligible Participants
Number analyzed (Participants) | 97
Participants
  Declined to hear about study | 22
  Agreed to hear about study: Consented | 52
  Agreed to hear about study: Did not consent | 23

3. Primary Outcome: Days to Hospital Day of Enrollment
Description: Days to hospital day of enrollment in relation to admission and discharge dates
Time Frame: approximately 3 months
Measure: Mean (Standard Error); unit: days
Arm/Group | Enhanced Opioid Stewardship Program | Standard of Care
Number analyzed (Participants) | 36 | 16
days | 9.66 (1.12) | 10.56 (2.30)
Statistical Analysis 1: Comparison: Enhanced Opioid Stewardship Program vs Standard of Care; Test type: Superiority; p = 0.69, t-test, 2 sided; Mean Difference (Net) = 0.89, 95% CI 2-sided [-3.67 to 5.46]

4. Primary Outcome: Number of Participants in the Intervention Group Who Were Able to Receive the Full Enhanced Opioid Stewardship Intervention
Description: Number of participants in the intervention group who were able to receive the full enhanced opioid stewardship intervention to determine retention
Time Frame: approximately 3 months
Population: Only participants in the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Opioid Stewardship Program
Number analyzed (Participants) | 36
Participants | 36

5. Primary Outcome: Number of Participants in Intervention Group Who Complete the Peri-discharge Evaluation.
Description: Number of participants in the intervention group who were able to complete the peri-discharge evaluation to determine retention.
Time Frame: approximately 3 months
Population: Only participants in the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Opioid Stewardship Program
Number analyzed (Participants) | 36
Participants
  Clinical outcomes provided | 36
  Self reported outcomes provided | 31

6. Primary Outcome: Number of Participants in Control Group Who Complete the Peri-discharge Evaluation.
Description: Number of participants in the control group who were able to complete the peri-discharge evaluation to determine retention.
Time Frame: approximately 3 months
Population: Only participants in the control group.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care
Number analyzed (Participants) | 16
Participants
  Clinical outcomes provided | 16
  Self-reported outcomes provided | 14

7. Secondary Outcome: Number of Guideline-based Care Elements in Use Considered Guideline Concordant Care With Opioids for Pain During Hospitalization.
Description: A a count of guideline-based care elements considered to be "best practices" for opioid stewardship in the setting of chronic pain will be collected during hospitalizations. These include ordering of alternative pain relief medications (e.g., acetaminophen), ordering of a bowel regimen, ordering of medication to treat opioid use disorder, order of urine toxicology screen, ordering of ECG for patients prescribed methadone, avoidance of co-prescriptions of benzodiazepines, and other associate "best care" practices. These metrics will be abstracted from the medical record. The number is out of a possible 12 recommendations- 12 would be the most recommendations a participant could have received.
Time Frame: approximately 4 months
Population: Only those in Enhanced Opioid Stewardship Program
Measure: Mean (Full Range); unit: Physician guideline-concordant recommend
Arm/Group | Enhanced Opioid Stewardship Program
Number analyzed (Participants) | 36
Physician guideline-concordant recommend | 4.4 [2 to 8]

8. Secondary Outcome: Change in Pain Intensity Measured by the Brief Pain Inventory - Severity
Description: The Brief Pain Inventory measures the intensity of pain, along with the degree to which the pain interferes with the everyday functioning of life. Scores range from 0 (no pain) to 10 (severe pain).
Time Frame: Baseline and 48 hours prior to discharge from hospital
Population: Participants with complete data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Enhanced Opioid Stewardship Program | Standard of Care
Number analyzed (Participants) | 30 | 14
score on a scale | -0.46 (0.26) | -0.23 (0.59)
Statistical Analysis 1: Comparison: Enhanced Opioid Stewardship Program vs Standard of Care; Test type: Superiority; p = 0.67, t-test, 2 sided; Mean Difference (Net) = 0.23, 95% CI 2-sided [-0.89 to 1.36]

9. Secondary Outcome: Change in Pain Intensity Measured by the Brief Pain Inventory - Interference
Description: The Brief Pain Inventory measures the intensity of pain, along with the degree to which the pain interferes with the everyday functioning of life. Scores range from 0 (no life interference) to 10 (complete interference).
Time Frame: Baseline and 48 hours prior to discharge from hospital
Population: Participants with complete data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Enhanced Opioid Stewardship Program | Standard of Care
Number analyzed (Participants) | 30 | 14
score on a scale | -1.21 (0.50) | -0.62 (0.64)
Statistical Analysis 1: Comparison: Enhanced Opioid Stewardship Program vs Standard of Care; Test type: Superiority; p = 0.50, t-test, 2 sided; Mean Difference (Net) = 0.59, 95% CI 2-sided [-1.16 to 2.34]

10. Secondary Outcome: Change in Depression Measured by the Patient Health Questionnaire
Description: The Patient Health Questionnaire measures Change in depression. Scores range from 0 (no depression) to 27 (severe depression).
Time Frame: Baseline and 48 hours prior to discharge from hospital
Population: Participants with complete data.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Enhanced Opioid Stewardship Program | Standard of Care
Number analyzed (Participants) | 30 | 14
score on a scale | -0.56 (0.38) | -0.35 (0.43)
Statistical Analysis 1: Comparison: Enhanced Opioid Stewardship Program vs Standard of Care; Test type: Superiority; p = 0.74, t-test, 2 sided; Mean Difference (Net) = 0.20, 95% CI 2-sided [-1.09 to 1.51]

11. Secondary Outcome: Patient Satisfaction Measured Using a Patient Satisfaction Survey
Description: Patient satisfaction will be measured using a Likert scale with scores ranging from a scale of 1-5 (1 not satisfied, 5 very satisfied). These data were not collected as part of the completed study.
Time Frame: 48 hours prior to discharge from hospital
Population: These data were not collected.
Arm/Group | Enhanced Opioid Stewardship Program | Standard of Care
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Count of Participants With Hospital Re-admissions at 30 Days After Hospitalization
Description: The Number of participants with hospital re-admissions at 30 days after hospitalization. Outcome was updated upon results entry.
Time Frame: up to 30 days post hospitalization
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Opioid Stewardship Program | Standard of Care
Number analyzed (Participants) | 36 | 16
Participants
  Readmission in 30 days: Yes | 14 | 4
  Readmission in 30 days: No | 22 | 12
Statistical Analysis 1: Comparison: Enhanced Opioid Stewardship Program vs Standard of Care; Test type: Superiority; p = 0.33, Chi-squared

13. Secondary Outcome: Count of Participants With Emergency Department Visit(s) at 30 Days After Hospitalization
Description: The count of participants with emergency department visits at 30 days after hospitalization. The outcome was updated when results were entered.
Time Frame: up to 30 days post hospitalization
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Opioid Stewardship Program | Standard of Care
Number analyzed (Participants) | 36 | 16
Participants
  ED Visit within 30 Days: Yes | 15 | 5
  ED Visit within 30 Days: No | 21 | 11
Statistical Analysis 1: Comparison: Enhanced Opioid Stewardship Program vs Standard of Care; Test type: Superiority; p = 0.47, Chi-squared

ADVERSE EVENTS:
Time Frame: Up to 4 months
Arm/Group | Enhanced Opioid Stewardship Program | Standard of Care
All-Cause Mortality (participants affected / at risk) | 1/36 | 0/16
Serious Adverse Events (participants affected / at risk) | 1/36 | 0/16
Other Adverse Events (participants affected / at risk) | 0/36 | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enhanced Opioid Stewardship Program (N=36) | Standard of Care (N=16)
Cardiorespiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-04): https://cdn.clinicaltrials.gov/large-docs/26/NCT05370326/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-04): https://cdn.clinicaltrials.gov/large-docs/26/NCT05370326/ICF_001.pdf